CLINICAL TRIAL: NCT01173354
Title: Essential Amino Acid Intake to Optimize Protein Anabolism in Elderly COPD Patients
Brief Title: EAA Intake to Optimize Protein Anabolism in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 105558
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Protein metabolism; Essential amino acid intake
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Excitatory Amino Acids; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD patients only (Experimental): Free balanced amino acid mixture or free essential amino acid mixture
  Interventions: Dietary Supplement: Free balanced amino acid mixture; Dietary Supplement: Free essential amino acid mixture

INTERVENTIONS:
Dietary Supplement: Free balanced amino acid mixture — 7 g free amino acids provided as a one time bolus, including 15 g carbohydrates. As part of the total amount of essential amino acids 24% is leucine.
  Other Names: 7 g AA (24% leucine of the EAA is leucine)
Dietary Supplement: Free essential amino acid mixture — 7 g free essential amino acids provided as a one time bolus, including 15 g carbohydrates. As part of the total amount of essential amino acids 40% is leucine.
  Other Names: 7 g EAA (including 40% leucine)

SUMMARY:
Weight loss commonly occurs in patients with chronic obstructive pulmonary disease (COPD), negatively influencing their quality of life, treatment response and survival. Loss of muscle protein is generally a central component of weight loss in COPD patients. Attempts to reverse muscle loss in COPD by supplying large amounts of protein or calories to these patients have been unsuccessful. Gains in muscle mass are difficult to achieve in COPD unless specific metabolic abnormalities are targeted. The investigators recently observed that alterations in protein metabolism are present in normal weight COPD patients. Elevated levels of protein synthesis and breakdown rates were found in this COPD group indicating that alterations are already present before muscle wasting occurs. Furthermore, reduced plasma essential amino acid (EAA) levels were observed in COPD patients. These reduced EAA plasma levels were significantly related with the presence of muscle wasting in COPD. Until now, limited research has been done examining protein metabolism and the response to feeding in patients with COPD. Previous studies support the concept of essential amino acids (EAA) as an anabolic stimulus in the young and elderly and in insulin resistant states. Until yet no information is present on the anabolic effects of EAA in elderly COPD patients.

It is therefore our hypothesis that a high-leucine essential amino acids mixture specifically designed to stimulate protein anabolism will target the metabolic alterations of COPD patients. In the present study, the acute effects of an EAA nutritional supplement on whole body, muscle and liver protein metabolism will be examined in COPD patients and compared to a supplement consisting of a balanced mixture of total amino acids. The principal endpoints will be the extent of stimulation of whole body protein synthesis as this is the principal mechanism by which either amino acid or protein intake causes muscle anabolism, and the reduction in endogenous protein breakdown. Both endpoints will be assessed by isotope methodology which is thought to be the reference method.

DETAILED DESCRIPTION:
In this study the investigators will test the following hypothesis: A high-leucine essential amino acid mixture (dose of 7.0 g EAA + 15 g carbohydrates) will stimulate protein anabolism to a greater extent than a standard balanced mixture of total (essential and non-essential) amino acids (dose of 6.7 g total AA + 15 g carbohydrates) in COPD patients. The principal endpoints will be the extent of stimulation of protein synthesis rate and the reduction in endogenous protein breakdown. The current project will provide information that will enable us to better understand the underlying metabolic mechanisms that regulate protein metabolism in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic airflow limitation, defined as measured forced expiratory volume in one second (FEV1) less than 70% of reference FEV1
* Shortness of breath on exertion
* Age 45 years and older
* Clinically stable condition and not suffering from respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the study
* Ability to lie in supine position for 6 hours

Exclusion Criteria:

* Established diagnosis of malignancy
* Presence of fever within the last 3 days
* Established diagnosis of Diabetes Mellitus
* Untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Recent myocardial infarction (less than 1 year)
* Use of long-term oral corticosteroids or short course of oral corticosteroids in the preceding month before enrollment
* Any other condition according to the PI or study physicians would interfere with proper conduct of the study / safety of the patient
* Failure to give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09-08 (Actual); Primary Completion 2012-02-17 (Actual); Study Completion 2012-02-17 (Actual)

PRIMARY OUTCOMES:
Net whole body protein synthesis rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement

SECONDARY OUTCOMES:
Whole body collagen breakdown rate | Up to 3 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Urea turnover rate | Up to 3 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Arginine turnover rate | Up to 3 years
  Measured in postabsorptive state
Muscle protein breakdown | Up to 3 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Amino acid kinetics | Up to 3 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Liver protein synthesis rate | Up to 3 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Resting Energy expenditure | Up to 3 years
  Measured in postabsorptive state
Insulin kinetics | Up to 3 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Glucose kinetics | Up to 3 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Fat-free mass | Up to 3 years
  Characterization of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Marielle PK Engelen, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951
- [Derived] Jonker R, Deutz NE, Erbland ML, Anderson PJ, Engelen MP. Alterations in whole-body arginine metabolism in chronic obstructive pulmonary disease. Am J Clin Nutr. 2016 Jun;103(6):1458-64. doi: 10.3945/ajcn.115.125187. Epub 2016 May 4. PMID 27146652